CLINICAL TRIAL: NCT02471677
Title: Corifollitropin Alfa (Elonva) Versus Follitropin Beta in High Responders: A Randomized Controlled Trial
Brief Title: Corifollitropin Alfa Versus Follitropin Beta in High Responders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eugonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: elonva_hyper-responders
Record Dates: First submitted 2015-06-08; First posted 2015-06-15 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Infertility
Keywords: Ovarian stimulation; corifollitropin alfa; GnRH antagonist protocol; high responders; follitropin beta
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Puregon (Active Comparator): Patients will undergo ovarian stimulation using daily injections of recombinant FSH (Puregon), as performed traditionally in IVF cycles
  Interventions: Drug: Puregon
- Elonva (Experimental): Patients will undergo ovarian stimulation using a single injection of corifollitropin alfa (Elonva)
  Interventions: Drug: Elonva

INTERVENTIONS:
Drug: Elonva — corifollitropin alfa (Elonva): a single injection 100 or 150 ug (depending on patient body weight) on Day 2/3 of menstrual cycle
  Other Names: corifollitropin alfa
  Arms: Elonva
Drug: Puregon — follitropin beta (Puregon): daily injections 150 IU from Day 2/3 of menstrual cycle until adequate follicle development is achieved
  Other Names: follitropin beta
  Arms: Puregon

SUMMARY:
The purpose of this randomized controlled trial (RCT) is to compare a single injection of corifollitropin-alfa versus daily injections of follitropin beta regarding the number of oocytes retrieved, hormonal profile and follicle development in patients with high response undergoing ovarian stimulation for in vitro fertilization treatment using a gonadotropin-releasing hormone (GnRH) antagonist protocol combined with GnRH agonist trigger and cryopreservation of all embryos.

DETAILED DESCRIPTION:
Corifollitropin alfa, a novel fusion protein lacking luteinizing hormone (LH) activity, has a longer elimination half-life and extended time to peak levels than recombinant follicle stimulating hormone (rFSH). A single injection of corifollitropin alfa may replace seven daily injections follitropin beta during the first week of ovarian stimulation, reducing patient discomfort.

The purpose of this RCT is to compare a single injection of corifollitropin-alfa versus daily injections of follitropin beta regarding the number of oocytes retrieved, as well as hormonal profile and follicle development in patients with high response undergoing ovarian stimulation for IVF using a GnRH antagonist protocol. In addition, incidence of unexpected ovarian hyperstimulation syndrome (OHSS) will be evaluated, although it is anticipated that GnRH agonist triggering will eliminate occurrence of the syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years
* Polycystic ovaries (PCO) or polycystic ovary syndrome (PCOS)
* no endometriotic cyst

Exclusion Criteria:

* Patients with poor response
* Patients using human chorionic gonadotropin (hCG) for triggering final oocyte maturation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | Day of oocyte retrieval (Day 0)

SECONDARY OUTCOMES:
Incidence of severe OHSS | up to 5 days post oocyte retrieval
Follicle development | Day of triggering final oocyte maturation = last day of ovarian stimulation (Day -2 prior to oocyte retrieval)
Fertilization rate | Day 1 after oocyte retrieval
Blastocyst formation rates | Day 5/6 after oocyte retrieval
Number of blastocysts cryopreserved | Day 5/6 after oocyte retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Trifon G Lainas, PhD, Study Director — Eugonia
Locations (1):
- Eugonia Unit of Assisted Reproduction, Athens, Greece

REFERENCES:
- [Background] Devroey P, Boostanfar R, Koper NP, Mannaerts BM, Ijzerman-Boon PC, Fauser BC; ENGAGE Investigators. A double-blind, non-inferiority RCT comparing corifollitropin alfa and recombinant FSH during the first seven days of ovarian stimulation using a GnRH antagonist protocol. Hum Reprod. 2009 Dec;24(12):3063-72. doi: 10.1093/humrep/dep291. Epub 2009 Aug 14. PMID 19684043
- [Background] Fauser BC, Alper MM, Ledger W, Schoolcraft WB, Zandvliet A, Mannaerts BM; Engage Investigators. Pharmacokinetics and follicular dynamics of corifollitropin alfa versus recombinant FSH during ovarian stimulation for IVF. Reprod Biomed Online. 2010 Nov;21(5):593-601. doi: 10.1016/j.rbmo.2010.06.032. Epub 2010 Jun 30. PMID 20843746
- [Background] Fauser BC, Mannaerts BM, Devroey P, Leader A, Boime I, Baird DT. Advances in recombinant DNA technology: corifollitropin alfa, a hybrid molecule with sustained follicle-stimulating activity and reduced injection frequency. Hum Reprod Update. 2009 May-Jun;15(3):309-21. doi: 10.1093/humupd/dmn065. Epub 2009 Jan 30. PMID 19182099